CLINICAL TRIAL: NCT01152008
Title: Evaluation Chez Des Sujets Sains d'Une Nouvelle Technique d'étude de la Microcirculation cutanée
Brief Title: Use of Laser Speckle to Study Cutaneous Blood Flow at Exercise in Healthy Subjects
Acronym: Speckle-move
Status: Completed | Type: Observational
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Other Study IDs: CHU P 2010-05
Record Dates: First submitted 2010-06-24; First posted 2010-06-29 (Estimated); Last update posted 2017-11-01 (Actual); Status verified 2010-07

CONDITIONS: Microcirculation
Keywords: Microcirculation; laser flowmetry; Skin; Physiology
MeSH Terms: interventions — Laser-Doppler Flowmetry

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- healthy volunteers
  Interventions: Other: tourniquet ischemia

INTERVENTIONS:
Other: tourniquet ischemia — Recording of cutaneous blood flow on the forearm at rest and during cycle exercise 50W before and following tourniquet ischemia
  Other Names: laser doppler flowmetry; Transcutaneous PO2; Near infra-red spectrometry

SUMMARY:
We aim to test the hypothesis that Laser speckle contrast imaging allows for the measurement of cutaneous blood flow during exercise.

DETAILED DESCRIPTION:
Ischemia and post occlusive reactive hyperhemia in the skin is tested in healthy normal subjects at rest and during cycle exercise.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers
* Affiliation to the French health system

Exclusion Criteria:

* Any disease or chronic treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: healthy volunteers
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2010-06; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Guillaume MAHE, MD, Principal Investigator — University Hospital in Angers
Locations (1):
- University Hospital, Angers, France

REFERENCES:
- [Derived] Mahe G, Haj-Yassin F, Rousseau P, Humeau A, Durand S, Leftheriotis G, Abraham P. Distance between laser head and skin does not influence skin blood flow values recorded by laser speckle imaging. Microvasc Res. 2011 Nov;82(3):439-42. doi: 10.1016/j.mvr.2011.06.014. Epub 2011 Jul 14. PMID 21784084